CLINICAL TRIAL: NCT07286929
Title: Evaluation of the Variation Over Time of Visuospatial Deficit in Patients With Parietal Lobe Glioma
Acronym: neGLIO
Status: Recruiting | Type: Observational
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Other Study IDs: neGLIO
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Glioma; Parietal Lobe Glioma; Visuspatial Deficit; Unilateral Spatial Neglect (USN)
Keywords: Visuospatial deficit; Glioma; Parietal Lobe; Neuropsychological assessment; Hemineglect
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of modern neurooncological surgery is to obtain maximum tumor resection while preserving neurological function. Parietal lobe gliomas often cause attention deficits (hemineglect) that are difficult to differentiate from other deficits. This study aims to evaluate the extent and variation over time of visuo-spatial deficits in patients undergoing surgical removal of parietal lobe gliomas. This will help characterize the cognitive profile of these patients to identify personalized treatment and rehabilitation paths.

DETAILED DESCRIPTION:
This is a single-centre, prospective, cross-sectional, observational study involving 40 patients with high- and low-grade parietal lobe glioma. The study investigates the prevalence of subjects who show a performance in cognitive visuo-spatial tests below the cut-off of the normative sample. It evaluates associations with patient-reported outcome measures (ADL, IADL), clinical-demographic aspects, radiological data (MRI), and histological/molecular data. Assessments occur at screening (pre-surgery), and at follow-up visits (3-4 months and 6 months post-surgery). Neuropsychological tests include Line Bisection, Bell and Letter Cancellation, Reading test, Apple Cancellation, and Fluff test.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years old
* Patients must understand the Italian Language
* Patients with suspected parietal lobe glioma

Exclusion Criteria:

* Tumor site other than parietal lobe.
* Patients who cannot undergo surgical resection (stereotactic/open biopsy).
* Patients who received a previous chemotherapy and/or radiotherapy treatment.
* Patients with a history of intracranial mass lesion or traumatic brain injury.
* Patients with a history of other CNS diseases (e.g., stroke, metastasis).
* Patients with diagnosis of neurodegenerative disease (i.e. Alzheimer's Disease, Frontotemporal Dementia, Parkinson's Disease, Lewy Body Dementia, Amyotrophic Lateral Sclerosis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected parietal lobe glioma
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in Visuospatial Deficit Prevalence | Baseline (pre-surgery), 3-4 months post-surgery, 6 months post-surgery.
  Prevalence of patients with a score below the cut-off in specific neuropsychological tests for visuo-spatial aspects (Line Bisection, Bell/Letter Cancellation, Apple Cancellation, Fluff Test) and the extent of change compared to baseline.

SECONDARY OUTCOMES:
Association with Radiological Data | Up to 6 months post-surgery
  Correlation between visuo-spatial deficit scores and MRI data (FLAIR volume, T1 contrast, necrosis, localization).
Association with Clinical-Demographic Data | Up to 6 months post-surgery.
  Correlation between visuo-spatial scores and hemispheric dominance, age, sex, and education.
Association with Performance Status | Time Frame: Up to 6 months post-surgery.
  Correlation between visuo-spatial scores and Karnofsky Performance Status (KPS).
Association with Histological/Molecular Data | Up to 6 months post-surgery.
  Correlation between visuo-spatial scores and tumor grade, histological and molecular features.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Di Meco, MD, Principal Investigator — Fondazione IRCCS Istituto Neurologico Carlo Besta
Locations (1):
- Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Italy

IPD SHARING:
Plan to Share IPD: No